CLINICAL TRIAL: NCT00318383
Title: A Phase 2, Multi-center, Randomized, Double-blinded, Placebo-controlled Study to Assess Efficacy of 3'-Aminomethylnicotine-P.Aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX) in Smokers Who Want to Quit Smoking
Brief Title: Efficacy of NicVAX in Smokers Who Want to Quit Smoking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Nabi Biopharmaceuticals (Industry)
Responsible Party: Matt Hohenboken, MD, PhD, Executive Dir., Clinical & Medical Affairs, Nabi Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nabi - 4512; 1R01DA017894-01A1 (NIH)
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-11

CONDITIONS: Smoking Cessation
Keywords: Vaccine; Immunogenicity; Randomized Controlled Trial
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): 200 mcg NicVAX in each of 4 doses
  Interventions: Biological: NicVAX conjugate vaccine
- 2 (Experimental): 200 mcg NicVAX in each of 5 doses
  Interventions: Biological: NicVAX conjugate vaccine
- 3 (Experimental): 400 mcg NicVAX in each of 4 doses
  Interventions: Biological: NicVAX conjugate vaccine
- 4 (Experimental): 400 mcg NicVAX in each of 5 doses
  Interventions: Biological: NicVAX conjugate vaccine
- 5 (Placebo Comparator): Placebo in 4 or 5 doses
  Interventions: Biological: Placebo
- 6 (Experimental): 200 mcg NicVAX formulation 2 in each of 5 doses
  Interventions: Biological: NicVAX conjugate vaccine

INTERVENTIONS:
Biological: NicVAX conjugate vaccine — 200 mcg or 400 mcg IM in 4 doses over 6 months; 200 mcg or 400 mcg IM in 5 doses over 6 months; 200 mcg (formulation 2) IM in 5 doses over 6 months; All are adsorbed onto Alhydrogel
  Other Names: 3'-aminomethylnicotine-rEPA conjugate vaccine
  Arms: 1; 2; 3; 4; 6
Biological: Placebo — Phosphate buffered saline and ALhydrogel of identical appearance to NicVAX; IM in 4 or 5 doses over 6 months
  Arms: 5

SUMMARY:
The purpose of this study is to determine whether vaccination with NicVAX will result in a higher continuous abstinence rate than vaccination with placebo in smokers who want to quit smoking. In addition, two different formulations and dosing schedules will be studied, to select the dose and dosing schedule which generates the highest level of anti-nicotine antibodies. The primary study period is 12 months, which was extended by amendment to include up to 2 years of observations.

DETAILED DESCRIPTION:
Cigarette smoking is responsible for over 400,000 (1 out of every 5) deaths in the United States each year. Most smokers are aware of the health consequences and want to quit, but have difficulty doing so. Only 3-5% of smokers who quit on their own are successful. Since the vast majority of those who attempt to quit will fail, the need for better approaches to smoking cessation is clear and urgent. A safe and effective means of blocking the effects of nicotine would be of considerable interest as a potential treatment for tobacco use. Vaccination to produce nicotine-specific antibodies may be viewed as an alternative method of blocking nicotine effects. Nicotine is a small molecule that does not elicit an immune response in animals of humans. In order for the immune system to respond to this hapten, nicotine can be combined or bound to a larger molecule in a unique manner so that an immune response is mounted against nicotine. Nabi Biopharmaceuticals has developed a conjugate vaccine (NicVAX) that consists of 3'-aminomethylnicotine bound to Pseudomonas aeruginosa exoprotein A, an exotoxin that has been made non-toxic by an amino acid deletion. Subjects will be randomized to one of four treatment groups.

Within each treatment group, 75 subjects will be randomized in a 2:1 ratio (NicVAX:Placebo), yielding a total of 50 active and 25 placebo subjects for each treatment group. There will be 12 subjects enrolled in a fifth open label arm to evaluate immunogenicity. A quit date will be set at the end of week 7 or at the end of week 5, depending on the dosing schedule. Continuous abstinence will be measured between the end of week 18 and the end of week 26.

ELIGIBILITY:
Inclusion Criteria:

* Smokes at least 15 cigarettes per day
* Wants to quit smoking
* Good general health
* Negative pregnancy test prior to study entry
* Carbon monoxide level greater than 10 ppm

Exclusion Criteria:

* Prior exposure to NicVAX or any other nicotine vaccine
* Known allergic reaction to alum or any of the components of the vaccine
* Use of steroids, immunosuppressive agents or other medication that might interfere with an immune response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Continuous smoking abstinence | 8 week interval (Weeks 19 to 26, inclusive, following the first vaccination)

SECONDARY OUTCOMES:
Point prevalence abstinence | at 12 months, and other time points; extended up to 24 months
Duration of smoking abstinence | at 6 and 12 months
Safety | 0-12 months, and extended up to 24 months
Numbers of cigarettes per day | Target quit day to 12 months
Cumulative number of cigarettes smoked | during weeks 18-26
Exhaled CO | at clinic visits
Urine cotinine | at clinic visits
Modified Minnesota Nicotine Withdrawal Questionnaire | weekly for 6 months, daily for 14 days after quit attempt
Cigarette Evaluation Questionnaire (a.k.a. Nabi Questionnaire) | weekly for 6 motnhs
Fagerstrom Test for Nicotine Dependence | baseline, weeks 26 and 52
serum anti-nicotine antibody concentrations by Elisa | periodic from baseline to month 12, extended to month 24

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hohenboken, MD, PhD, Study Director — Nabi Biopharmaceuticals
Locations (9):
- United States (9):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California, San Francisco, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Department of Public & Community Health, College Park, Maryland
  - Tobacco Research Center, Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oregon Health & Science University, Portland, Oregon
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Fahim RE, Kessler PD, Fuller SA, Kalnik MW. Nicotine vaccines. CNS Neurol Disord Drug Targets. 2011 Dec;10(8):905-15. doi: 10.2174/187152711799219343. PMID 22229310
- [Derived] Hatsukami DK, Jorenby DE, Gonzales D, Rigotti NA, Glover ED, Oncken CA, Tashkin DP, Reus VI, Akhavain RC, Fahim RE, Kessler PD, Niknian M, Kalnik MW, Rennard SI. Immunogenicity and smoking-cessation outcomes for a novel nicotine immunotherapeutic. Clin Pharmacol Ther. 2011 Mar;89(3):392-9. doi: 10.1038/clpt.2010.317. Epub 2011 Jan 26. PMID 21270788